CLINICAL TRIAL: NCT04020679
Title: A Hybrid Implementation-effectiveness Stepped Wedge Cluster Randomised Controlled Trial to Determine the Effectiveness of the Goals of Care Initiative
Brief Title: The Goals of Care Initiative
Acronym: GOCI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18_CPCR_17
Record Dates: First submitted 2019-07-10; First posted 2019-07-16 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Decision-Making Oncology; Chemotherapy Effect

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Cluster Randomised Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Participants will not receive GOCI materials
- Intervention (Experimental): Participants will receive GOCI materials and clinicians will receive training.
  Interventions: Behavioral: Goals of Care Initiative

INTERVENTIONS:
Behavioral: Goals of Care Initiative — Can-GUIDE will provide videos on a number of SDM topics including interviews with patients and clinicians discussing patient involvement in SDM and how goal conversations can inform the decision making process. Furthermore, there will be instructional videos on how to complete the Goal conversations sheet. Accompanying the videos will be interactive elements which will help users consider the types of questions that they wish to ask their clinical teams. The goal conversation sheet allows patients to list their goals and priorities that they wish to bring up in the consultation with their clinical teams. The Goals of Care (GOC) tool is a communication aid for clinicians to summarise goals of care discussions such as those facilitated by the goals conversation sheet. The completed tool will then be logged onto the Electronic Patient Record (EPR) and is then disseminated to other HCPs involved in the patients care.
  Other Names: Can-GUIDE
  Arms: Intervention

SUMMARY:
A single site hybrid implement-evaluation stepped wedge cluster randomised controlled trial in which cancer cluster groups (lung, colorectal, breast, renal, ovarian, upper GI & sarcoma) are randomised sequentially to initiate the Goals of Care Initiative into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing, or being considered for, systemic treatment from one of the cluster teams.
* 18+ years.
* Able to give written consent.
* Able to understand verbal and written English.

Exclusion Criteria:

• Patient is not being considered for Systemic Anti-Cancer Treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
SDM-Q-9 | Immediately following intervention
  Patient involvement in decision making will be measured using the SDM-Q-9 questionnaire. The questionnaire contains nine items with respondents scoring on a six point scale (0 represents completely disagree to 5 which represents completely disagree) how much they agree with the presented statement. The highest score attainable, 45, represents the highest level of perceived Shared Decision Making and 0 represents no perceived involvement in Shared Decision Making.
Decision Conflict Scale | Immediately following intervention
  Patient satisfaction with decision and overall decision conflict will be measured using the Ottawa Decisional Conflict Scale. The scale consists of 16 items with patients scoring themselves on a five point scale (0, Strongly Agree - 4, Strongly Disagree). The scale includes five subscales: uncertainty, support, values, informed, effective decision.
  The total score and subscale scores are calculated by dividing the sum of the items by the number of items within that subscale and multiplying by twenty five (scored range from 0 to 100; 0 score indicates no decisional conflict, 100 indicates extremely high decisional conflict). This scale evaluates the quality of decision as outlined within internationally recognised guidelines to establish the effectiveness of decision aids. Furthermore, some of the subscales address evaluating the quality of the decision process (feeling informed about the options, clarity of values).

SECONDARY OUTCOMES:
Decision Self Efficacy Scale | Immediately following intervention, then at 6 weeks and 12 weeks.
  A patient's ability to make a decision about treatment (or decision self-efficacy) will be measured using the Ottawa Decision Self-Efficacy scale. The scale consists of 11 items where patients score themselves on a five point scale (0, not at all confident - 4, Very confident); high score indicates greater decision self-efficacy. The total score provides a global rating of self confidence in the patient's ability to engage with decision making regarding their treatment. The total score is calculated by summing the 11 items, dividing by 11 and then multiply by 25.
EQ-5D-5L | Immediately following intervention, then at 6 weeks and 12 weeks.
  EQ-5D is a standardised instrument for use as a measure of health outcome and it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care as well as in population health surveys. The EuroQoL 5-level version (EQ-5D-5L) will be assessed to provide a preference based measure of health-related quality-of-life which will enable us to calculate a quality adjusted life-year (QALY) for use in the cost-effectiveness analysis. The preference weights to estimate utility values and QALYs will be those recommended by NICE at the time of data analysis.
  Participants are asked to choose a statement which best relates to their current experience relating to the following health domains: mobility, self-care, ability to carry out usual activities, pain/discomfort, anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Janelle Yorke, PhD, Principal Investigator — University of Manchester
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided